CLINICAL TRIAL: NCT02643303
Title: A Phase 1/2 Study of In Situ Vaccination With Tremelimumab and IV Durvalumab (MEDI4736) Plus the Toll-like Receptor Agonist Poly-ICLC in Subjects With Advanced, Measurable, Biopsy-accessible Cancers
Brief Title: A Study of Tremelimumab and IV Durvalumab Plus Poly-ICLC in Subjects With Biopsy-accessible Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: MedImmune LLC (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2014-011
Record Dates: First submitted 2015-12-18; First posted 2015-12-31 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Breast Cancer; Sarcoma; Merkel Cell Carcinoma; Cutaneous T-Cell Lymphoma; Melanoma; Renal Cancer; Bladder Cancer; Prostate Cancer; Testicular Cancer; Solid Tumor
Keywords: Durvalumab; MEDI4736; Tremelimumab; Poly-ICLC; Hiltonol®; Breast Cancer; Melanoma; In Situ; CTLA-4 Antibody; PD-L1 Antibody; TLR3 Agonist; CTCL; Imfinzi®
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Sarcoma; Carcinoma, Merkel Cell; Lymphoma, T-Cell, Cutaneous; Melanoma; Kidney Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Testicular Neoplasms | interventions — durvalumab; tremelimumab; poly ICLC

STUDY DESIGN:
Intervention Model Description: In Phase 1, Cohort 1A was opened first and after the safety of durvalumab and poly-ICLC was demonstrated, Cohorts 1B and 1C were open in parallel. In Phase 2, all tumor types were opened in parallel, and subjects included in Cohort 1C were included and reported in their respective tumor type in Phase 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1, Cohort 1A (Experimental): Subjects received durvalumab (1500 mg IV every 4 weeks [Q4W] for 12 cycles). Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Poly-ICLC
- Phase 1, Cohort 1B (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (75 mg IV Q4W for the first 4 cycles).
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Sarcoma (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Merkel Cell Carcinoma (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Cutaneous T-cell Lymphoma (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Genitourinary Cancers with Accessible Metastases (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC
- Cohort 1C + Phase 2; Solid Tumors with Accessible Masses (Experimental): Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Poly-ICLC

INTERVENTIONS:
Drug: Durvalumab
  Other Names: MEDI4736; Imfinzi®
Drug: Tremelimumab
  Arms: Cohort 1C + Phase 2; Cutaneous T-cell Lymphoma; Cohort 1C + Phase 2; Genitourinary Cancers with Accessible Metastases; Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma; Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer; Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies; Cohort 1C + Phase 2; Merkel Cell Carcinoma; Cohort 1C + Phase 2; Sarcoma; Cohort 1C + Phase 2; Solid Tumors with Accessible Masses; Phase 1, Cohort 1B
Drug: Poly-ICLC
  Other Names: Hiltonol®

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study of the CTLA-4 antibody, tremelimumab, and the PD-L1 antibody, durvalumab (MEDI4736), in combination with the tumor microenvironment (TME) modulator poly-ICLC, a TLR3 agonist, in subjects with advanced, measurable, biopsy-accessible cancers.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/2 study of the cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody, tremelimumab, and the programmed cell death ligand-1 (PD-L1) antibody, durvalumab (MEDI4736), in combination with the tumor microenvironment (TME) modulator poly-ICLC, a toll-like receptor 3 (TLR3) agonist, in subjects with advanced, measurable, biopsy-accessible cancers. Subjects will receive intratumoral and intramuscular (IM) administration of poly-ICLC and intravenous (IV) administration of durvalumab, together with either IV or intratumoral administration of tremelimumab. The study will be conducted in 2 phases.

Phase 1: There will be enrollment to 3 subject cohorts in Phase 1, with staggered initiation of enrollment.

* Cohort 1A: IV Durvalumab + Intratumoral/IM Poly-ICLC. After safety is demonstrated in the first 3-6 subjects in Cohort 1A, Cohorts 1B and 1C will open to enrollment.
* Cohort 1B: IV Durvalumab + IV Tremelimumab + Intratumoral/IM Poly-ICLC.
* Cohort 1C: IV Durvalumab + Intratumoral Tremelimumab + Intratumoral/IM Poly-ICLC.

Phase 2: Upon determination of the recommended combination dose in Cohort 1C, up to 66 evaluable subjects will be treated in Phase 2. Up to 6 subjects will be initially enrolled by tumor type (head and neck squamous cell carcinoma, locally recurrent or metastatic breast cancer, sarcoma, Merkel cell carcinoma, cutaneous T-cell lymphoma, melanoma after failure of available therapies, genitourinary cancers and solid tumors with accessible metastases). Subjects enrolled in Cohort 1C will be included in Phase 2 in the applicable tumor type. Data from all subjects in each Phase 2 tumor type will be reviewed for safety/efficacy to select up to 3 tumor types that demonstrate an efficacy signal, defined as at least 1 of 6 subjects within a tumor type who achieve a partial response (PR) or complete response (CR) by immune-related RECIST (irRECIST) or RECIST 1.1, or stable disease (SD) for at least 6 months. Up to 6 additional subjects in each of the selected tumor types may be enrolled in the expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologic confirmation of advanced, biopsy-accessible, measurable cancers of the following histologies:

   * Non-viral-associated head and neck squamous cell carcinoma (HNSCC) or human papillomavirus (HPV)-associated HNSCC after failure of prior therapy
   * Locally recurrent or metastatic breast cancer
   * Sarcoma
   * Merkel Cell Carcinoma (MCC)
   * Cutaneous T cell Lymphoma (CTCL)
   * Melanoma after failure of available therapies
   * Genitourinary (GU) cancers with accessible metastases (e.g., bladder, renal)
   * Any solid tumors with masses that are accessible
2. Subjects with measurable disease, must have at least 2 lesions (1 measurable lesion and 1 biopsy/injectable lesion, which does not need to be measurable).
3. Any number of prior systemic therapies.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Laboratory parameters for vital functions should be in the normal range or not clinically significant.

Exclusion Criteria:

1. Prior treatment with combination CTLA-4 and PD-1/PD-L1 blockade, with the exception of subjects with melanoma.
2. Participants may not have been treated intratumorally with poly-ICLC.
3. Subjects with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any active brain metastases, or, within 6 months of the first date of treatment on this study, history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage.
4. Active, suspected or prior documented autoimmune disease, clinically significant cardiovascular disease or clinically uncontrolled hypertension.
5. History of pneumonitis or interstitial lung disease or any unresolved immune-related adverse events following prior biological therapy.
6. Other malignancy within 2 years prior to entry into the study, except for those treated with surgical therapy only (e.g., localized low-grade cervical or prostate cancers).
7. Subjects with clinical symptoms or signs of gastrointestinal obstruction and/or who require drainage gastrostomy tube and/or parenteral hydration or nutrition.
8. Known immunodeficiency or HIV, Hepatitis B, or Hepatitis C positivity. Antibody to Hepatitis B or C without evidence of active infection may be allowed.
9. History of severe allergic reactions to any unknown allergens or any components of the study drugs.
10. Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
11. History of allogeneic organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, Jr., MD, Study Chair — University of Virginia; Nina Bhardwaj, MD, PhD, Study Chair — Tisch Cancer Institute Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - Research Facility, Atlanta, Georgia
  - Research Facility, Lebanon, New Hampshire
  - Research Facility, Buffalo, New York
  - Research Facility, New York, New York
  - Research Facility, Cleveland, Ohio
  - Research Facility, Toledo, Ohio
  - Research Facility, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Bohnsack O, Hoos A, Ludajic K. Adaptation of the immune related response criteria: irRECIST. Ann Oncol. 2014 Sep;25(suppl 4):iv361-iv72 [Abstract 4958]. doi: 10.1093/annonc/mdu342.23.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 subjects were enrolled and 56 treated with at least one dose of study treatment.
Pre-assignment Details: The Phase 1 Cohort 1C dosing regimen was used in Phase 2 without any dose modifications. As indicated in the protocol, the subjects enrolled in Cohort 1C are included in the appropriate Phase 2 cohort based on tumor type. For this reason, Cohort 1C is not presented separately.
Groups:
- Phase 1, Cohort 1A: Subjects received durvalumab (1500 mg IV every 4 weeks [Q4W] for 12 cycles). Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Durvalumab
  Poly-ICLC
- Phase 1, Cohort 1B: Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (75 mg IV Q4W for the first 4 cycles).
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Durvalumab
  Tremelimumab
  Poly-ICLC
- Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma; Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer; Cohort 1C + Phase 2; Sarcoma; Cohort 1C + Phase 2; Merkel Cell Carcinoma; Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies; Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases; Cohort 1C + Phase 2; Solid Tumors With Accessible Masses: Subjects received durvalumab (1500 mg IV Q4W for 12 cycles) and tremelimumab (10 mg) intratumorally on days 1, 8, and 15 of Cycle 1, days 1 and 15 of Cycle 2 and day 1 of Cycles 3 and 4.
  Poly-ICLC (1 mg) was administered intratumorally on days 1, 3, 5, 8, 10 and 15 and intramuscularly on days 17, 22, and 24 of Cycle 1 as well as intramuscularly on days 1, 3, 8, 10, 15, 17, 22 and 24 of Cycle 2 and on days 1 and 4 of Cycle 3.
  Durvalumab
  Tremelimumab
  Poly-ICLC
Period: Overall Study
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Started (Subjects who started treatment.) | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7
Completed (Subjects who completed 12 cycles of treatment.) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Not Completed | 4 | 5 | 1 | 13 | 7 | 4 | 9 | 3 | 7
Not completed — Progressive Disease | 4 | 4 | 1 | 12 | 6 | 4 | 8 | 2 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses | Total
Number analyzed (Participants) | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7 | 56
Age, Continuous [Median (Full Range); unit: years] | 52.5 [37 to 70] | 55 [26 to 69] | 66 [66 to 66] | 59 [39 to 71] | 51 [21 to 68] | 66 [46 to 71] | 64 [34 to 84] | 54 [45 to 55] | 58 [31 to 80] | 58 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 0 | 15 | 2 | 1 | 6 | 0 | 4 | 36
  Male | 1 | 0 | 1 | 0 | 5 | 3 | 4 | 3 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 5 | 1 | 14 | 7 | 4 | 10 | 3 | 6 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 7
  White | 4 | 5 | 1 | 11 | 5 | 3 | 7 | 3 | 6 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7 | 56
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    ECOG PS 0 | 2 | 0 | 0 | 6 | 4 | 2 | 4 | 1 | 4 | 23
    ECOG PS 1 | 2 | 5 | 1 | 9 | 3 | 2 | 6 | 2 | 3 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) were reported based on clinical laboratory tests, vital signs, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent was signed through 90 days after the last dose of study treatment. Treatment-emergent AEs were those that occurred or worsened after administration of the first dose of study treatment.
Time Frame: up to 15 months
Population: All subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7
Participants
  Number of Subjects with TEAEs | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7
  Number of Subjects with Treatment-Related TEAEs (TRAEs) | 4 | 4 | 1 | 13 | 6 | 3 | 10 | 1 | 7
  Number of Subjects with Serious TRAEs | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Subjects with Dose-Limiting Toxicities (DLTs) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Subjects who Died on Study | 0 | 2 | 0 | 3 | 1 | 1 | 1 | 2 | 0

2. Primary Outcome: Number of Subjects With Best Overall Tumor Response by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 21 days before the first dose of study treatment), and in Cycles 4, 7, 9 and 11, when a subject discontinued treatment prematurely and 28 days after the last dose of study treatment. Per irRECIST, measurable lesions were categorized as follows: Complete Response (irCR): Complete disappearance of all target lesions; Partial Response (irPR): ≥ 30% decrease from baseline in the Total Measured Tumor Burden (TMTB); Progressive Disease (irPD): ≥ 20% increase from nadir in Total Measured Tumor Burden (TMTB); Stable Disease (irSD): not meeting above criteria.
Time Frame: up to 15 months
Population: All subjects who had at least one dose of study medication and one baseline and at least one post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 4 | 1 | 14 | 7 | 4 | 9 | 2 | 6
Participants
  irCR | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  irPR | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  irSD | 2 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 3
  irPD | 1 | 4 | 1 | 9 | 6 | 4 | 6 | 2 | 3

3. Secondary Outcome: Median Progression-free Survival (PFS) by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) as Estimated Using the Kaplan-Meier Method
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 21 days before the first dose of study treatment), and in Cycles 4, 7, 9 and 11, when a subject discontinued treatment prematurely and 28 days after the last dose of study treatment.
  PFS was measured from the date of the first dose of study treatment to the date of earliest disease progression according to irRECIST or to the date of death, if disease progression did not occur. Per irRECIST, Progressive Disease (irPD) was defined as a ≥ 20% increase from nadir in the Total Measured Tumor Burden (TMTB).
Time Frame: up to 15 months
Population: All subjects who had at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7
days | 157 [82 to NA] — The upper limit of the confidence interval was not estimable due to the small number of events. | 44 [21 to NA] — The upper limit of the confidence interval was not estimable due to the small number of events. | 85 [NA to NA] — The upper and lower limits of the confidence interval were not estimable due to the small number of events. | 85 [42 to 225] | 44 [9 to 83] | 68 [37 to NA] — The upper limit of the confidence interval was not estimable due to the small number of events. | 82 [26 to 127] | 43 [24 to NA] — The upper limit of the confidence interval was not estimable due to the small number of events. | 84 [37 to NA] — The upper limit of the confidence interval was not estimable due to the small number of events.

4. Secondary Outcome: Overall Disease Control Rate as Measured by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 21 days before the first dose of study treatment), and in Cycles 4, 7, 9 and 11, when a subject discontinued treatment prematurely and 28 days after the last dose of study treatment. Per irRECIST, measurable lesions were categorized as follows: Complete Response (irCR): Complete disappearance of all target lesions; Partial Response (irPR): ≥ 30% decrease from baseline in the Total Measurable Tumor Burden (TMTB); Progressive Disease (irPD): ≥ 20% increase from nadir in Total Measured Tumor Burden (TMTB); Stable Disease (irSD): not meeting above criteria.
  Overall Disease Control Rate was defined as the percentage of subjects who had irSD for at least 6 months, or irPR or irCR over a period of at least 4 weeks. Subjects who dropped out prior to meeting the responder criteria were considered non-responders.
Time Frame: Up to 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 4 | 1 | 14 | 7 | 4 | 9 | 2 | 6
Participants | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Subjects With Best Overall Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 21 days before the first dose of study treatment), and in Cycles 4, 7, 9 and 11, when a subject discontinued treatment prematurely and 28 days after the last dose of study treatment. Per RECIST 1.1, target lesions are categorized as follows: Complete Response (CR): disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions or presence of new lesions; Stable Disease (SD): small changes that did not meet above criteria.
Time Frame: up to 13 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 4 | 1 | 14 | 7 | 4 | 9 | 2 | 6
Participants
  CR | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  SD | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 3
  PD | 1 | 4 | 1 | 9 | 7 | 4 | 6 | 2 | 3

6. Secondary Outcome: Median PFS by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as Estimated Using the Kaplan-Meier Method
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 21 days before the first dose of study treatment), and in Cycles 4, 7, 9 and 11, when a subject discontinued treatment prematurely and 28 days after the last dose of study treatment.
  PFS was measured from the date of the first dose of study treatment to the date of earliest disease progression according to RECIST 1.1 or to the date of death, if disease progression did not occur. Per RECIST 1.1, Progressive disease (PD) was defined as a ≥ 20% increase in the sum of the longest diameter of target lesions or the presence of new lesions.
Time Frame: Up to 15 months
Population: All subjects who had at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7
days | 157 [82 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 44 [21 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 85 [NA to NA] — Upper and lower limits of confidence interval were not estimable due to the small number of events. | 85 [42 to 225] | 44 [9 to 83] | 68 [37 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 82 [26 to 127] | 43 [24 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 84 [37 to NA] — Upper limit of confidence interval was not estimable due to the small number of events.

7. Secondary Outcome: Overall Disease Control Rate as Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 21 days before the first dose of study treatment), and in Cycles 4, 7, 9 and 11, when a subject discontinued treatment prematurely and 28 days after the last dose of study treatment. Per RECIST 1.1, target lesions are categorized as follows: Complete Response (CR): disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions or presence of new lesions; Stable Disease (SD): small changes that did not meet above criteria.
  Overall Disease Control Rate was defined as the percentage of subjects who had SD for at least 6 months, or PR or CR over a period of at least 4 weeks. Subjects who dropped out prior to meeting the responder criteria were considered non-responders.
Time Frame: up to 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 4 | 1 | 14 | 7 | 4 | 9 | 2 | 6
Participants | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Median Overall Survival (OS) as Estimated Using the Kaplan-Meier Method
Description: After completion of treatment, all subjects were followed for survival every 3 months for 2 years after completion of treatment; then every 6 months until 5 years from study entry; then yearly until 10 years from study entry. OS was measured from the date of the first dose of study treatment to the date of death or last follow-up. Subjects lost to follow-up were censored on the date when they were last known to be alive. Per protocol amendment 6.0, all post study follow-up for the collection of survival data was discontinued as of February 28, 2022. The last collection of survival data was on February 23, 2022.
Time Frame: up to 5 years
Population: All subjects that had at least one study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
Number analyzed (Participants) | 4 | 5 | 1 | 15 | 7 | 4 | 10 | 3 | 7
days | 1238 [266 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 129 [26 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 338 [NA to NA] — Upper and lower limits of confidence interval were not estimable due to the small number of events. | 326 [68 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 300 [64 to 370] | 224 [74 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 202 [51 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 43 [39 to NA] — Upper limit of confidence interval was not estimable due to the small number of events. | 565 [264 to NA] — Upper limit of confidence interval was not estimable due to the small number of events.

ADVERSE EVENTS:
Time Frame: All AEs occurring between the signing of informed consent and the off-study date (i.e., through 90 days after the last dose of study treatment) are documented, regardless of the causal relationship to study drug). AEs that occur or worsen in severity after the first dose of study treatment are considered treatment emergent (i.e., TEAEs). All-cause mortality includes all deaths which were reported up to 5 years.
Description: AE documentation includes onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Phase 1, Cohort 1A | Phase 1, Cohort 1B | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer | Cohort 1C + Phase 2; Sarcoma | Cohort 1C + Phase 2; Merkel Cell Carcinoma | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses
All-Cause Mortality (participants affected / at risk) | 3/4 | 5/5 | 1/1 | 9/15 | 6/7 | 4/4 | 6/10 | 3/3 | 6/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/5 | 0/1 | 4/15 | 3/7 | 2/4 | 3/10 | 2/3 | 2/7
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 1/1 | 15/15 | 7/7 | 4/4 | 10/10 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Cohort 1A (N=4) | Phase 1, Cohort 1B (N=5) | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma (N=1) | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer (N=15) | Cohort 1C + Phase 2; Sarcoma (N=7) | Cohort 1C + Phase 2; Merkel Cell Carcinoma (N=4) | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies (N=10) | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases (N=3) | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Cohort 1A (N=4) | Phase 1, Cohort 1B (N=5) | Cohort 1C + Phase 2; Head + Neck Squamous Cell Carcinoma (N=1) | Cohort 1C + Phase 2; Locally Recurrent or Metastatic Breast Cancer (N=15) | Cohort 1C + Phase 2; Sarcoma (N=7) | Cohort 1C + Phase 2; Merkel Cell Carcinoma (N=4) | Cohort 1C + Phase 2; Melanoma After Failure of Available Therapies (N=10) | Cohort 1C + Phase 2; Genitourinary Cancers With Accessible Metastases (N=3) | Cohort 1C + Phase 2; Solid Tumors With Accessible Masses (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2 | 3 | 1 | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Excess cerumen production (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 7 | 0 | 0 | 2 | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 1 | 4 | 5 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 2 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 1 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 1 | 7 | 1 | 3 | 8 | 3 | 5
Chills (General disorders) | 1 | 0 | 0 | 8 | 2 | 2 | 4 | 0 | 0
Injection site pain (General disorders) | 1 | 2 | 1 | 7 | 3 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 3 | 4 | 2 | 2 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 1 | 2
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Injection site reaction (General disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localized oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood cortisol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 5 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 3 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 4 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tumour exudation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 3 | 2 | 2 | 4 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 5 | 0 | 2 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Delerium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 2 | 1 | 3 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess drainage (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02643303/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT02643303/SAP_001.pdf